CLINICAL TRIAL: NCT00561652
Title: Education/Exercise and Chiropractic for Chronic Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Northwestern Health Sciences University (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B5027-R
Record Dates: First submitted 2007-11-19; First posted 2007-11-21 (Estimated); Results first posted 2015-02-10 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-01

CONDITIONS: Low Back Pain
Keywords: Low back pain; Chiropractic; Exercise; Veterans
MeSH Terms: conditions — Low Back Pain; Motor Activity | interventions — Educational Status; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Education + exercise (Active Comparator): Education was provided in four, 1-hour sessions to improve patients' understanding of their back problem, reduce unwarranted concern about serious outcomes, & empower them to maintain normal activities & reduce risk of future back problems. Patients were taught that recovery depends on moving & restoring normal function & fitness. Patients were shown stretching & strengthening exercises to perform daily at home to enhance mobility & increase trunk endurance while minimizing spinal load. At follow-up, therapists reviewed exercise form & adherence. Participants allocated to no chiropractic care also were scheduled for 10 weekly 10-15 minute sessions to equalize provider attention vs. the group also receiving chiropractic care & not to provide education, exercise instruction, or therapy.
  Interventions: Behavioral: Education & Exercise
- Education + exercise + chiropractic (Experimental): In addition to education & exercise, all participants in this arm will be assigned chiropractic treatment. A minimum of 4 & up to 12 treatments will be provided over 6 weeks, based on patient response (i.e. treatments stopped if symptoms resolve). Each treatment visit will last 10-20 minutes. After 6 weeks, if the treating chiropractor determined that the patient's LBP was continuing to improve but hadn't reached therapy goals defined at baseline, the patient could receive up to 12 additional treatments over the next 6 weeks. Chiropractic treatment was delivered following standardized protocols. Treatment consisted of manual therapies, including SMT and mobilization techniques, with the assistance of light soft tissue techniques as indicated to facilitate the SMT.
  Interventions: Behavioral: Education & Exercise; Procedure: Chiropractic treatment (plus Education & Exercise)

INTERVENTIONS:
Behavioral: Education & Exercise — Education & Exercise
Procedure: Chiropractic treatment (plus Education & Exercise) — Chiropractic treatment (plus Education & Exercise)
  Arms: Education + exercise + chiropractic

SUMMARY:
As a needed first step prior to a planned full-scale RCT, in order to assess the feasibility of the RCT and refine its design and protocols, we will perform a pilot study with the following objectives:1.To assess whether enough veterans with chronic LBP can be identified, meet eligibility criteria and be randomized to demonstrate that recruitment for a planned full-scale RCT is feasible. 2.To assess whether veterans with chronic LBP will adhere to protocol interventions per study protocol. 3.To assess whether veterans with chronic LBP will complete data collection per study protocol. 4.To obtain estimates of effect sizes and the corresponding standard errors of the primary efficacy outcome measures to estimate the required sample size of a planned full-scale RCT.

DETAILED DESCRIPTION:
Chronic low back pain (LBP) is associated with poor health, lower quality of life, high costs, and is highly prevalent in veterans. Both chiropractic care and exercise have modestly reduced pain and/or improved function in randomized controlled trials (RCTs) of patients with chronic LBP. However, effects may not apply similarly to all populations. For example, there are no RCT data on chiropractic care for older (age >70) patients with chronic LBP, though with increased spinal arthritis, comorbidities and frailty, such patients may require modified chiropractic techniques and likely differ in response to chiropractic treatment. While a recent systematic review of RCTs predicted that a home exercise program that was individualized, high-dose, therapist-directed, and incorporated stretching and strengthening would be a meaningful treatment for chronic LBP, it also could provide a robust comparison group for other chronic LBP treatments. The combination of such a regimen and chiropractic care is predicted to have additive benefits for chronic LBP but this premise hasn't been directly tested. To further our aim of improving the health of chronic LBP patients, we plan an RCT in veterans with chronic LBP, to compare the effectiveness, cost-effectiveness and cost-utility of a tailored education/exercise (E/E) intervention alone vs. E/E plus chiropractic care. The demographics and medical complexity of the veteran population provide a great opportunity to test the appropriate role of chiropractic care for such patients with chronic LBP and to advance chronic LBP research and clinicalcare.

Subjects will be recruited primarily from patients attending Minneapolis VAMC clinics with complaints of chronic LBP. Thirty eligible veterans will be randomized to E/E alone vs. E/E plus chiropractic care. All participants will receive E/E instruction in four 1-hr individual sessions over 8 weeks, including an individually designed, high dose, therapist-directed home exercise program. Chiropractic care will be delivered by chiropractors and follow standard protocols, with up to 12 sessions over 12 weeks. Participants randomized to E/E alone also will attend 10 weekly "time and attention" visits so that their contact with providers is comparable to that received by participants who also receive chiropractic care. Each "time and attention" session involved a 5 minute exam, 5 minutes of hot pack application to the low back, and 5 minutes of light massage to the low back. During these visits, participants did not receive SMT, mobilization or other active chiropractic treatment. The recruitment goal is to generate the potential to randomize 6-10 participants/month. Recruitment feasibility will be assessed by tracking the number of patients who make initial inquiries, undergo screening and in-clinic evaluation, and are randomized. Further, reasons for nonparticipation and disqualification will be examined and described. Participant adherence to interventions will be defined as completing >3 of 4 education sessions, >20 hrs of home exercise, and >80% of recommended chiropractic visits or nonchiropractic follow-up exam/interviews. Adherence with clinic visits will be assessed with provider treatment logs. Home exercise compliance will be tracked by questionnaire. Participant adherence to data collection will be defined as >90% follow-up rates at each time point and assessed by tracking questionnaire completion rates. Descriptive data for the distributions of the primary and main secondary efficacy outcome measures will be used to calculate sample size and generate power tables for the full-scale trial.

ELIGIBILITY:
Inclusion Criteria:

* Veterans enrolled to receive VA medical care
* Current low back pain episode present > 6 weeks.
* LBP pain score > 3 on scale of 0-10.
* LBP classified using the Quebec Task Force (QTF) system as types 1-4 respectively, patients with LBP, stiffness or tenderness, without radiation; with radiation proximal to knee; with radiation distal to knee; or with radiation and >2 abnormal neurological exam findings.
* No change in past month in prescription medications affecting musculoskeletal pain.

Exclusion Criteria:

* Low back pain classified as QTF type 5-11
* Progressive neurologic deficits due to nerve root or spinal cord compression, including symptoms/signs of cauda equina syndrome.
* Previous lumbar spine surgery, by history and/or screening spine radiograph.
* Acute vertebral fracture, by history and spine radiograph
* Self-reported ongoing LBP treatment by other healthcare providers other than stable prescription medications affecting musculoskeletal pain.
* Infectious and noninfectious inflammatory destructive spine tissue changes, by spine radiograph
* Self-reported pending/current litigation pertaining to back pain, including workers compensation claims; or pending evaluation of VA service connected rating related to back pain.
* Clinically significant chronic inflammatory spinal arthritis
* Self-reported pregnancy
* Self-reported current substance abuse
* History of bleeding disorder
* Known arterial aneurysm near LBP area
* Possible/confirmed spinal/vertebral infection, by history and spine radiograph
* Primary or metastatic vertebral malignancy, by history and spine radiograph

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-04; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard A. Fink, MD MPH, Principal Investigator — Minneapolis Veterans Affairs Medical Center
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Veterans were recruited between 1/2008 & 3/2009 at the Minneapolis VA, with flyers given to patients presenting to Primary Care, Physical Therapy & Orthopedics clinics with low back pain; recruitment posters; & mailings to patients previously diagnosed with back pain.
Pre-assignment Details: 1075 were offered initial phone screening, 71 completed further in-clinic screening, & 30 were randomized. Participants were randomly assigned to treatment groups at the time of enrollment with no wash out, run-in, or transition between enrollment and group assignment. No enrolled participants were excluded from the trial before group assignment.
Groups:
- Arm 1: Education plus exercise
- Arm 2: Chiropractic treatment plus education plus exercise
Period: Overall Study
Arm/Group | Arm 1 | Arm 2
Started | 10 | 20
Completed | 10 | 19
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 10 | 20 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 12 | 19
  >=65 years | 3 | 8 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 9 | 17 | 26
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaskan Native | 0 | 0 | 0
  Asian or Pacific Islander | 0 | 1 | 1
  Nonhispanic Black | 0 | 0 | 0
  Hispanic | 1 | 1 | 2
  Nonhispanic White | 9 | 18 | 27
Region of Enrollment [Number; unit: participants]
  United States | 10 | 20 | 30

OUTCOME MEASURES:

1. Other Pre Specified Outcome: Participant Adherence With Chiropractic Visits
Description: Number of participants who completed at least 12 chiropractic visits.
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 0 | 20
participants |  | 18

2. Primary Outcome: Participant Adherence With Education + Exercise Visits
Description: Number of participants completing at least 3 of 4 education + exercise visits
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 10 | 20
participants | 9 | 19

3. Other Pre Specified Outcome: Participant Adherence With "Time and Attention" Visits
Description: Number of participants who completed at least 8 of 10 "time and attention" visits. Note that only arm 1 (nonchiropractic arm) receives "time and attention" visits.
Time Frame: 12 weeks
Population: Only arm 1 received "time and attention" visits as their purpose was to balance the chiropractor provider contact time received by arm 2 participants.
Measure: Number; unit: participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 10 | 0
participants | 1 |

4. Other Pre Specified Outcome: Participant Adherence With Prescribed Home Exercise
Description: Number of participants who completed at least 20 hours of home exercise
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 10 | 20
participants | 2 | 10

5. Other Pre Specified Outcome: Participant Adherence With Week 6 Follow-up Questionnaire
Description: Number of participants who completed their week 6 follow-up questionnaire
Time Frame: 6 weeks
Measure: Number; unit: participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 10 | 20
participants | 8 | 16

6. Other Pre Specified Outcome: Participant Adherence With Week 12 Follow-up Questionnaire
Description: Number of participants who completed their week 12 follow-up questionnaire
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 10 | 20
participants | 9 | 18

7. Other Pre Specified Outcome: Participant Adherence With Week 26 Follow-up Questionnaire
Description: Number of participants who completed week 26 follow-up questionnaire
Time Frame: 26 weeks
Measure: Number; unit: participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 10 | 20
participants | 6 | 15

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Participants were administered a questionnaire asking whether they had or hadn't experienced each of 7 possible adverse effects at each chiropractic and exercise therapist visit.
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/20
Other Adverse Events (participants affected / at risk) | 6/10 | 18/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (N=10) | Arm 2 (N=20)
Increase in low back pain (Musculoskeletal and connective tissue disorders) | 6 | 16
New leg pain (Musculoskeletal and connective tissue disorders) | 0 | 7
Different pain (General disorders) | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No